CLINICAL TRIAL: NCT04465773
Title: Pupillary Diameter Variations in Response to Tetanic Stimulations of Incremental Intensities in Patients Under Propofol-remifentanil TCI
Brief Title: Pupillary Response to Incremental Tetanic Stimulations Under Propofol-remifentanil TCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pr Isabelle CONSTANT (Other)
Responsible Party: Sponsor-Investigator, Pr Isabelle CONSTANT, Professor, Hôpital Armand Trousseau
Organization: Hôpital Armand Trousseau (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pupillo propofol remi stim
Record Dates: First submitted 2016-01-12; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Pain
Keywords: general anesthesia
MeSH Terms: conditions — Pain | interventions — Anesthesia, General; Propofol; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pupillometry (Experimental): General anesthesia for scheduled gynecological surgery Propofol target concentration adjusted to maintain bispectral index between 45 and 55 for 10 minutes Remifentanil target concentration 1 ng/ml for 10 minutes Tetanic stimulations of 10-20-30-40-50-60 milliamps (5 seconds per stimulation, 2 minutes between stimulations) Continuous pupillometry VideoAlgesiGraph
  Interventions: Procedure: general anesthesia for scheduled gynecological surgery; Drug: Propofol; Drug: Remifentanil, Ultiva®; Procedure: tetanic stimulations; Device: VideoAlgesiGraph

INTERVENTIONS:
Procedure: general anesthesia for scheduled gynecological surgery
Drug: Propofol — continuous infusion, target concentration adjusted to maintain bispectral index between 45 and 55
Drug: Remifentanil, Ultiva® — continuous infusion, target concentration 1 ng/ml
Procedure: tetanic stimulations — 10-20-30-40-50-60 milliamps, 5 seconds, 100 Hertz 2 minutes between stimulations delivered via the standard neuromuscular blocking agents monitor
Device: VideoAlgesiGraph — non invasive infrared camera placed in front of the left eye of the patients during the study period, connected to a laptop. No part of the device touches the eye.
  Other Names: VideoAlgesiGraph, Synapsis (TM), Marseille, France

SUMMARY:
In patients under standardized steady-state general anesthesia, 6 tetanic stimulations of incremental intensities were applied to the patients. Pupillary dilation in response to these stimulations was recorded.

DETAILED DESCRIPTION:
The aim of the study was to investigate a possible correlation between the intensity of a nociceptive stimulus and the magnitude of pupillary reflex dilation in patients anesthetized with propofol and remifentanil target-controlled infusion.

Anesthetic protocol: 10 minutes of steady-state general anesthesia (before extubation during a scheduled gynecological surgery) with remifentanil target concentration of 1 ng/ml, and propofol target concentration adjusted to maintain bispectral index between 45 and 55.

Study period: 6 tetanic stimulations of incremental intensities were applied to the patients: 10, 20, 30, 40, 50, 60 milliamps Pupillary dilation in response to these stimulations was recorded.

Then, propofol and remifentanil infusions were discontinued, and patients were extubated.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled gynecological surgery requiring general anesthesia and orotracheal intubation
* written informed consent

Exclusion Criteria:

* ophthalmic disease
* neurologic disease
* preoperative chronic pain or pain medication
* medication interfering with autonomous nervous system (beta blockers, alpha agonists, metoclopramide, droperidol, atropine, catecholamines)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pupillary diameter | 5 seconds before tetanic stimulation
  as measured by VideoAlgesiGraph, in mm
Pupillary diameter | 1 minute after tetanic stimulation
  as measured by VideoAlgesiGraph, in mm

SECONDARY OUTCOMES:
Heart rate | 5 seconds before tetanic stimulation
  as measured by the standard cardioscope
Heart rate | 1 minute after tetanic stimulation
  as measured by the standard cardioscope

CONTACTS AND LOCATIONS:
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France